CLINICAL TRIAL: NCT04613908
Title: Efficacy of Conventional Rehabilitation, Transcutaneous Electro Nerve Stimulation or Early Mobilization to Reverse the Acquired Weakness of the Intensive Care Unit: Single Blind Controlled Clinical Trial
Brief Title: Efficacy of Different Treatments for the Intensive Care Unit Acquired Weakness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Nacional Profesor Alejandro Posadas (Other)
Responsible Party: Principal Investigator, Ladislao Diaz Ballve, Principal Investigator, Hospital Nacional Profesor Alejandro Posadas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02-2018
Record Dates: First submitted 2018-06-21; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Muscle Weakness; Rehabilitation
Keywords: Intensive Care Unit Acquired Weakness; Electric Stimulation Therapy; Early Mobility; Standard Rehabilitation Treatment
MeSH Terms: conditions — Muscle Weakness | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: 3 Groups Group 1 (GR-STD) received the standard or usual rehabilitation treatment used in our ICU as intervention.
  Group 2 (GR-NMES) received neuro muscular electro stimulation sessions in addition to the standard treatment.
  Group 3 (GR-EM) received an early mobilization protocol as intervention.
Who Masked: Outcomes Assessor
Masking Description: the person in charge of performing the statistical analysis was blind, by coding the interventions in the database.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard care or usual rehabilitation (Active Comparator): It will consist of the usual treatment performed by the intensive care physiotherapist, it will be applied every day that the study lasts.
  Interventions: Other: standard care or usual rehabilitation
- neuro muscular electro stimulation (Experimental): They received 5 sessions per week (except weekends) of neuromuscular electrostimulation of 30 minutes duration. Also, every day that the study is carried out in the morning and in the afternoon, the subjects will receive the usual treatment performed by the intensive care physiotherapist.
  Interventions: Device: neuro muscular electro stimulation
- early mobilization protocol (Experimental): Throughout the duration of the study, an early mobilization protocol will be applied to apply a specific treatment based on different levels of treatment for each subject of the group; It differs from the usual procedure in protocolized progression according to the objectives reached by the patient, unlike the usual treatment, where the progression is in accordance with the clinical criteria of the treatment professional.
  Interventions: Other: Early Mobilization protocol

INTERVENTIONS:
Device: neuro muscular electro stimulation — We used a commercial equipment of electro stimulation with a pulse width of 300 micro seconds, a frequency of 50 Hz, with symmetrical balanced biphasic rectangular wave and with an intensity of up to 80 milliampere.
  Other Names: DEMAX® model Quatrum Duo
  Arms: neuro muscular electro stimulation
Other: Early Mobilization protocol — The protocol consisted in applying a specific treatment based on different levels of treatment to each subject. Admission to them was carried out according to the maximum capacity of each subject, the conditions of each level being the following:
  * Level 1: MRC (shoulder) <3 + MRC <3 (hip).
  * Level 2: MRC (shoulder) ≥ 3 + MRC (hip) <3.
  * Level 3: MRC (shoulder) ≥ 3 + MRC (hip) ≥ 3 + sitting on the edge of the bed without assistance (minimum 15 minutes).
  * Level 4: Standing without assistance and walking with or without assistance.
  Arms: early mobilization protocol
Other: standard care or usual rehabilitation — routine, non-protocolized rehabilitation treatment performed by the physiotherapist assigned to intensive care
  Arms: standard care or usual rehabilitation

SUMMARY:
Experimental study that has how to compare the efficacy between conventional rehabilitation, transcutaneous electrostimulation or early mobilization to reduce the time needed to reverse the muscle weakness evaluated by the muscle strength scale of the MRC in patients with a clinical diagnosis of intensive care unit acquired weakness in the (ICUAW).The ambit of realization is a medical-surgical ICU of a general acute hospital (26 beds). A randomized controlled, uni-centric design was used. The interventions are divided into three groups namely; group 1 (control group) receiving standard or usual rehabilitation (GR-STD); group 2 receives transcutaneous electrostimulation (GR-TEE) and group 3 that consists of an early mobilization protocol (GR-EM). The main outcome variable of the study is the time, in days and sessions of treatment, to reverse the ICUAW.

DETAILED DESCRIPTION:
Study hypothesis: the time to revert the intensive care unit acquired weakness is less when applying an early mobilization protocol or transcutaneous electro-nervous stimulation compared with the usual or standard rehabilitative treatment.

Ethical considerations: The research protocol was presented and approved by both the Ethics Committee and the Teaching and Research Committee of our institution. The informed consent of each subject included in the study was obtained.

Sample size and study power: a sample size was defined in 18 subjects (6 subjects per intervention group). The estimation of the sample was calculated for a one-way ANOVA where a minimum difference of 2 sessions was established between the treatments, assuming a standard deviation of 1.8 sessions, an alpha error of 5% and a power of 80%.

Statistical methods: the numerical variables will be presented as mean and standard deviation or median and interquartile range according to the presented distribution. The categorical variables will be presented by frequency and percentage.

For the comparison of continuous variables, Student's t test for independent samples or the Mann-Whitney U test will be used according to the presented distribution and for the categorical variables the Chi² test or the Fisher exact test will be used according to the conformation of the crossed table. The Shapiro-Wilk test will be used to evaluate whether the distribution presented by the numerical variables fits a normal distribution. Equality of variances was assessed by the Levene´s test.

The comparison of the time to reach an smuscle strength scale of the MRC ≥ 48 between the groups with different interventions will be used the one-way ANOVA test or the Kruskal-Wallis test as appropriate. For post hoc analysis, the pairs-comparison test of Games-Hollew or Dunn's-Bonferroni will be used for ANOVA or Kruskal-Wallis, respectively, when they reach statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* subjects over 18 years of age,
* admitted to the ICU who have received invasive mechanical ventilation for a period longer than 24 hours
* clinical diagnosis of ICUAW (MRC-mss <48 measured over two consecutive days).

Exclusion Criteria:

* subjects who presented a body mass index> 35 (kg/height x height)
* presence of edema that prevents the realization of NMES at the time of diagnosis of ICUAW (assessed by the absence of visible contraction
* pregnant women
* subjects with pacemakers
* subjects with injury of the central and / or peripheral nervous system (with motor sequelae)
* previous neuromuscular disease
* limitation of the movement of any extremity due to orthopedic or traumatological causes
* presence of a previous cognitive disorder that impedes the understanding of rehabilitation interventions
* a value of the index of Barthel less than 35 points at admission
* subjets who refused to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
days needs to revert ICUAW | 3 months
  Number of days until reaching a value of the MRC-mss ≥ 48 points.
Sessions needs to revert ICUAW | 3 months
  Number of sessions until reaching a value of the MRC-mss ≥ 48 points.

CONTACTS AND LOCATIONS:
Overall Officials: Ladislao P Diaz Ballve, Principal Investigator — Hospital Nacional Posadas

IPD SHARING:
Plan to Share IPD: No